CLINICAL TRIAL: NCT06212635
Title: Novel Biomarkers for Evaluation of Hemostasis and Inflammation in Liver Cirrhosis
Brief Title: Hemostasis in Liver Cirrhosis and Hepatocellular Cancer
Acronym: HELICS
Status: Recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00316200610
Record Dates: First submitted 2023-02-22; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2023-02

CONDITIONS: Hemostasis in Decompensated Liver Cirrhosis; Inflammation in Decompensated Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Hemostasis assays, inflammation assays, DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Non-acute decompensated liver círrhosis: Refractory ascites, low grade encephalopathy but manages to stay at home and only come in ofr check-ups.
  Interventions: Diagnostic Test: T-TAS
- Acute decompensated liver cirrhosis: Acute event causing further decompensation and the need for in-patient care
  Interventions: Diagnostic Test: T-TAS
- Acute on chronic liver failure: ACLF 1-3 accordic to criterias established through the Cannonic study.
  Interventions: Diagnostic Test: T-TAS
- Controls: Healthy individuals
  Interventions: Diagnostic Test: T-TAS

INTERVENTIONS:
Diagnostic Test: T-TAS — Blood test, laboratory assays
  Other Names: Quantra; OHP

SUMMARY:
Evaluating hemostasis in decompensated liver cirrhosis with novel hemostatic assays.

DETAILED DESCRIPTION:
The rebalanced hemostasis in liver cirrhosis is vulnerable and patients are prone to both bleeding and thrombosis. There are today no gold standard for evaluating the hemostasis and we will evaluate novel methods for this.

ELIGIBILITY:
Inclusion Criteria:

* Patients with decompensated liver cirrhosis
* 18 years or older.
* Healthy individuals 18 years or older will serve as controls.

Exclusion Criteria:

* • Extrahepatic malignancy or recurrence of such within the last year.

  * Diagnosis of non-cirrhotic coagulopathy, coagulation disorder or thrombophilia prior to inclusion.
  * Diagnosis of hematological disease such as hematologic malignancies, non-cirrhotic thrombocytopenia or thrombocytosis, Polycytemia Vera, hemoglobinopathies
  * Previous liver transplantation.
  * Transfusions the last 7 days.
  * Treatment with platelet inhibitors or anticoagulant except for prophylactic dosage of LMWH. If a prophylactic dose of LMWH has been used study sampling with addition of antiFXa must be taken >12 hours after the last injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 40 patients each with NAD, AD and ACF and 30 healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Differences in laboratory values between groupstests | up to 5 years
  Laboratory values of novel hemostasis tests TTAS, Quantra and OHP correlated to Rotem, TG and conventional coagulation assays. All tests have differnet values.
Correlation between systemic inflammation and hemostasis measured by novel assays | uo to 7 years
  Correlation between systemic inflammation measured by cytokines, NETs and ECV and hemostasis measured by novel assays as in outcome 1

SECONDARY OUTCOMES:
Number of participant with bleeding | Up to 7 years
  Bleeding defined according to ISTH
Number of participants with Thrombosis | Up to 7 years
  Splanchnic or non-splanchnic thrombosis
Number of participants that die | Up to 7 years
Number of participant going to transplant | Up to 7 years
  Number of patients getting a transplant, acute, subacute or according to waiting list

CONTACTS AND LOCATIONS:
Overall Officials: Maria Magnusson, MD, PhD, Principal Investigator — Region Stockholm, Karolinska Institute
Locations (1):
- Karolinska University Hospital, Stockholm, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: Undecided